CLINICAL TRIAL: NCT01215565
Title: A Multicenter National Phase II Open Study Coupled With Translational Assessment of Biomarkers Predictive of Response to Sunitinib in Patients With Advanced/Inoperable Fibrolamellar Hepatocellular Carcinoma.
Brief Title: Study of Sunitinib in Patients With Advanced/Inoperable Fibrolamellar Carcinoma
Acronym: Fibrolam
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of inclusion
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P070134; 2008-003423-23 (EudraCT Number)
Record Dates: First submitted 2010-09-24; First posted 2010-10-06 (Estimated); Last update posted 2014-03-13 (Estimated); Status verified 2014-03

CONDITIONS: Hepatocellular Carcinoma; Fibrolamellar Hepatocellular Carcinoma
Keywords: Carcinoma, Hepatocellular; Carcinoma; Fibrosis; Liver Neoplasms; Pathologic Processes; Digestive System Neoplasms; Neoplasms by Site; Neoplasms; Liver Diseases; Adenocarcinoma; Neoplasms, Glandular and Epithelial; Neoplasms by Histologic Type; Sunitinib; Antineoplastic Agents; Therapeutic Uses; Pharmacologic Actions; Angiogenesis Inhibitors; Angiogenesis Modulating Agents; Growth Substances; Physiological Effects of Drugs; Growth Inhibitors
MeSH Terms: conditions — Carcinoma, Hepatocellular; Fibrolamellar hepatocellular carcinoma; Carcinoma; Fibrosis; Liver Neoplasms; Pathologic Processes; Digestive System Neoplasms; Neoplasms by Site; Neoplasms; Liver Diseases; Adenocarcinoma; Neoplasms, Glandular and Epithelial; Neoplasms by Histologic Type | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- patient treated (Experimental): patient who receive sunitinib
  Interventions: Drug: Sutent

INTERVENTIONS:
Drug: Sutent — Sunitinib 50mg/day (per os) for 6 cycles duration of one cycle = 6 weeks (4 weeks of treatment over 6 weeks)

SUMMARY:
The purpose of this study is to evaluate the antitumor activity of sunitinib in patients with advanced/inoperable fibrolamellar hepatocellular carcinoma.

Rationale: Sunitinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor

DETAILED DESCRIPTION:
Fibrolamellar hepatocellular carcinoma is variant rare of hepatocellular carcinoma witch distinct clinical, histological and prognostic features from conventional hepatocellular carcinoma. This entity typically occurs in young adults with no underlying hepatitis or cirrhosis. Surgical resections could be proposed in some referral centers and this in cases of localized tumors. However, in cases of postoperative recurrence, "salvage" resection is not often possible. Overall prognosis remains poor, because of its primary chemoresistance and early recurrence of metastasis.

Sunitinib (SUTENT) is a potent tyrosine kinase inhibitor, with double antiangiogenic and antitumor activity, targeting multiple receptors as VEGF-R, PDGF-R, KIT and FLT3.

Since 2006, Sunitinib has been approved to treat advanced kidney cancer also called advanced renal cell carcinoma (a typically chemoresistant disease for which there no active treatment was available).

Several targets of sunitinib are overexpressed hepatocellular carcinoma lines as shown in the Literature review and pathological studies.

Otherwise, the overexpression of PDGFR and VEGFR correlates with recurrence and invasion in HCC. Finally, sunitinib showed an interesting antitumor activity in patients with conventional advanced HCC.

Thereby, it seems important to study how well the sunitinib, a potent antitumor and antiangiogenic agent, works in treating patients with advanced or inoperable fibrolamellar hepatocellular carcinoma especially, this setting lacks effective therapies. Furthermore, it seems urgent to conduct translational research and assessment to identify predictive biomarkers of response.

In this study, orally sunitinib at dosed of 50 mg daily will be administrated to patients for 4 weeks, followed by 2 weeks of wash out. This administration schedule is based on the phase I study of sunitinib.

ELIGIBILITY:
Inclusion Criteria:

* Fibrolamellar hepatocellular carcinoma histopathologically proven
* Inoperable/advanced (Tumor recurrence inoperable or metastatic with no surgical indication).
* Available Tumor tissue for analysis(biopsy or surgical specimen)
* Performance status WHO ≤ 2.
* Adequate organ function :

  * Hematology (absolute neutrophil count equal or superior to 1,5 x 10*9/l , platelet equal or superior to 100 x 10*9/l),
  * clearance of creatinine > 60 ml/min),
  * AST/ALT ≤ 5 N, PAL ≤ 5 N, total bilirubin ≤ 2N.

Exclusion Criteria:

* Hypersensitivity to sunitinib.
* Contraindication to sunitinib, including uncontrolled hypertension, medical history of cerebrovascular accident, unstable cardiac pathology despite optimal medical therapy (myocardial infarction within the 6 months prior to study drug administration, severe/unstable angina ), active hemorrhagic syndrome or concomitant treatment with anticoagulants.
* Any severe acute or chronic co-morbid that may compromise to comply with study participation : uncontrolled infection, symptomatic congestive heart failure, liver disturbance, chronic renal failure, active gastro-duodenal ulcer (nonexhaustive list)
* Known brain metastases.
* Diagnosis of any second malignancy within the last 3 years, except for basal cell or squamous cell skin cancer, or in situ carcinoma of the cervix uteri
* Current treatment on another clinical trial.
* Prior treatment with an investigational agent within 4 weeks
* Patient on i.v bisphosphonate therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2009-10; Primary Completion 2011-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Objective response | 1 year
  to evaluate the objective response according to RECIST Criteria 1.1

SECONDARY OUTCOMES:
Objective response | 1 year
  to evaluate objective response to sunitinib according to secondary radiological criteria (evaluation on CT scan of: tumor density, % of tumor necrosis and tumor vascularisation)
Overall survival | 6 months and 1 year
Progression-Free survival | 6 months and 1 year
Biomarkers of response | 1 year
  to evaluate the correlation between biomarkers expression and objective response so sunitinib
Biomarkers of radiological response | 1 year
  to evaluate the correlation between biomarkers expression and secondary radiological criteria (significant decrease of tumor density on CT scan, formation of significant intratumor necrosis, significant decrease of tumoral vascularisation using of perfusion software

CONTACTS AND LOCATIONS:
Overall Officials: Sandrine Faivre, Professor, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hôpital Beaujon, Clichy, Hauts de Seine, France